CLINICAL TRIAL: NCT04828239
Title: Institutional Review Board of Kuang Tien General Hospital
Brief Title: Acupuncture Versus Laser Acupuncture for Carpal Tunnel Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kuang Tien General Hospital (Other)
Responsible Party: Principal Investigator, Li-Feng Lin, TCM department, Kuang Tien General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KTGH10946
Record Dates: First submitted 2021-03-24; First posted 2021-04-02 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Carpal Tunnel Syndrome
Keywords: laser acupuncture; Carpal Tunnel Syndrome; manual acupuncture
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: The recruited patients were randomly divided into two groups of ''Laser Acupuncture Group'' and ''Manual Acupuncture Group"
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Laser Acupuncture Group (Experimental): Acupuncture point: PC-6 and PC-7 laser pen is vertical to the points and with the pen at a distance of 0.5- cm from the skin., every point is treated for 1 min administrated over 4 weeks (2 sessions/wk)
  Interventions: Device: laser acupuncture
- Manual Acupuncture Group (Active Comparator): Acupuncture point: PC-6 and PC-7 Responses elicited: de qi sensation Manual: twirling with lifting-thrusting method stimulation Needles retained for 30 min Needle type: C&G, gauge and size: 0.25x40mm
  Interventions: Other: acupuncture
- Sham Laser Acupuncture Group (Sham Comparator): Acupuncture point: PC-6 and PC-7 Sham laser pen is vertical to the points and with the pen at a distance of 0.5- cm from the skin., every point is treated for 1 min administrated over 4 weeks (2 sessions/wk)
  Interventions: Device: Sham laser acupuncture

INTERVENTIONS:
Device: laser acupuncture — 400 mW, near-infrared, continuous wavelength, 810 nm. about 24J/cm2
  Other Names: RJ-LASER, Germany
  Arms: Laser Acupuncture Group
Other: acupuncture — Needle type: C&G, gauge and size: 0.25x40mm
  Arms: Manual Acupuncture Group
Device: Sham laser acupuncture — This laser pen is the same device with a red light was pasted on the acu-points in the same way, using the same protocol as for the active laser stimulation, but the laser apparatus was not switched on.
  Other Names: RJ-LASER, Germany
  Arms: Sham Laser Acupuncture Group

SUMMARY:
Carpal tunnel syndrome (CTS) results from the entrapment neuropathy of median nerve at the wrist, and most cases are idiopathic. So far, there are many treatments were developed (Surgical decompression, local injection of steroids, Wrist splints) but they are not fully satisfactory, other treatment modalities need to be further evaluated.

Both Acupuncture and laser acupuncture treatments for CTS have been reported. However, those studies still lack associated evidence to evaluate the efficacy of acupuncture and laser acupuncture.

The object of the study is to investigate the efficacy of acupuncture compared with laser acupuncture in patients with mild-to-moderate carpal tunnel syndrome (CTS). Nerve conduction studies (NCS) and global symptom score (GSS) assessment will apply to measure objective changes in this randomized, controlled study.

DETAILED DESCRIPTION:
Both manual acupuncture and laser acupuncture treatments for CTS have been reported.

Laser acupuncture (LA) is defined as the stimulation of traditional acupuncture points by using low-level intensity. Its a noninvasive treatment than acupuncture for those patients had the potential risk for infection or people involving pain or fear of needles. So far, previous studies still lack associated evidence about comparisons between laser acupuncture and manual acupuncture to evaluate their efficacy. So the investigators would like to compare the efficacy of acupuncture treatment with laser acupuncture (LA) treatment in patients with idiopathic, mild-to-moderate carpal tunnel syndrome (CTS)

ELIGIBILITY:
Inclusion Criteria:

CTS diagnosis was based on the presence of at least one of the following symptoms

1. numbness, tingling pain, or paresthesia in the median nerve distribution
2. precipitation of these symptoms by repetitive hand activities, which could be relieved by resting, rubbing, and shaking the hand
3. nocturnal awakening by such sensory symptoms.
4. The diagnosis was often supported by a positive Tinel sign Confirmed by the presence of one or more of the following standard electrophysiologic criteria

(1) prolonged distal motor latency (DML) to the abductor pollicis brevis (APB) (abnormal Z4.7 ms, stimulation over the wrist, 8 cm proximal to the active electrode) (2) prolonged antidromic distal sensory latency (DSL) to the second digit (abnormal Z3.1 ms;stimulation over the wrist, 14 cm proximal to the active electrode) (3) prolonged antidromic wrist-palm sensory nerve conduction velocity (W-P SNCV) at a distance of 8 cm (W-P SNCV, abnormal <45 m/s).9-

Exclusion Criteria:

1. Symptoms occurring less than 3 months before the study (to exclude patients who might have spontaneous resolution of symptoms)
2. severe CTS that had progressed to visible muscle atrophy
3. clinical or electrophysiologic evidence of accompanying conditions that could mimic CTS or interfere with its evaluation, such as cervical radiculopathy, proximal median neuropathy, or significant polyneuropathy
4. evidence of obvious underlying etiologic factors of CTS such as diabetes mellitus, rheumatoid arthritis, hypothyroidism (acromegaly), pregnancy, alcohol abuse or drug usage (steroids or drugs acting through the central nervous system), and suspected malignancy or inflammation or autoimmune disease documented as underlying causes of CTS
5. cognitive impairment interfering with the subject's ability to follow instructions and describe symptoms

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-03-10 (Actual); Primary Completion 2022-05-20 (Estimated); Study Completion 2022-06-20 (Estimated)

PRIMARY OUTCOMES:
Global symptom score | Change from Baseline GSS at 2 weeks
  rated symptoms(Pain ,Numbness, paresthesia, Nocturnal awakening) from 0(no symptoms) to 10 (very severe symptoms)
Global symptom score | Change from Baseline GSS at 4 weeks
  rated symptoms(Pain ,Numbness, paresthesia, Nocturnal awakening) from 0(no symptoms) to 10 (very severe symptoms)

SECONDARY OUTCOMES:
Nerve conduction studies | Change from Baseline nerve conduction studies (NCS) at 4 weeks
  calculate the median nerve transduction speed

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Pai Yang, PhD, Principal Investigator — Kuang Tien Genreal Hospital
Locations (1):
- Kuang Tien Genreal Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No